CLINICAL TRIAL: NCT04523012
Title: Seroprevalence of SARS-CoV-2 Infection in Patients With HIV Infection
Brief Title: COVID-19 and HIV Patients
Acronym: COCOVIH
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 013
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A venous blood sample will be taken as part of routine care for HIV: on D0 (a 6 ml tube will be collected), M6 (a 6 ml tube will be collected) and M12 (a 6 ml tube will be collected) during the recommended assessments for HIV management as part of routine care.
  On inclusion, after information and collection of the non-objection, a tube of blood (D0) will be collected during the assessment of the HIV infection and a control to determine the appearance or persistence of the antibodies will be done at M6 and M12 always as part of the assessment of HIV infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV patients: On inclusion, after information and collection of the non-objection, a blood sample (D0) will be taken during the assessment of the HIV infection (no unplanned sample will be taken) and a control to determine the appearance or the Persistence of antibodies will be made at M6 and M12 always as part of the assessment of HIV infection.
  Interventions: Other: Seroprevalence of SARS-CoV-2 infection in patients with HIV infection

INTERVENTIONS:
Other: Seroprevalence of SARS-CoV-2 infection in patients with HIV infection — On inclusion, after information and collection of the non-objection, a blood sample (D0) will be taken during the assessment of the HIV infection (no unplanned sample will be taken) and a control to determine the appearance or the Persistence of antibodies will be made at M6 and M12 always as part of the assessment of HIV infection.

SUMMARY:
As of May 26, 2020, 5,508,904 confirmed cases (145,279 in France) of COVID-19 and 346,508 deaths (28,457 in France) have been reported since December 8, 2019 worldwide. The rapid increase in the number of cases in our territory caused France to pass to level 3 of the epidemic on March 14, 2020.

The natural history of this disease is still poorly understood, particularly in patients infected with HIV, patients considered to be at higher risk for severe forms.

Knowing the seroprevalence in the population of people living with HIV will make it possible to better understand the Covid infection in immunocompromised patients, know the percentage of immunization and the persistence or not of the antibodies over time, specify the protective nature or not of these antibodies detected.

DETAILED DESCRIPTION:
To date, very little data is available in HIV-infected patients with Sars-Cov-2 infection. Only 11 cases of HIV patients with confirmed Sars-Cov-2 infection have been described in the literature. These patients are under 50 years of age, HIV infection with a controlled viral load in 8/11, 2 patients with a severe course requiring administration of tociluzumab, including one patient who died. In addition, the management of these HIV patients is not codified. Some authors have changed antiretroviral therapy to a protease inhibitor such as lopinavir or darunavir because of encouraging results in vitro but debated in patients. This clearly illustrates the disparity of approaches and the lack of data in this patient population.

Knowing the seroprevalence in the population of people living with HIV will allow us to better understand the Covid-19 infection in immunocompromised patients, know the percentage of immunization and the persistence or not of the antibodies over time as well as their unknown neutralizing effect. until now. No data exist on seroprevalence in the HIV population.

Serological tests can detect the immune response to COVID-19 in serum. Studies to date have shown seroconversion typically within two weeks of symptom onset, with notable differences depending on the studies, techniques and epitopes of the antigens chosen to detect the antibodies. A study which showed that the seropositivity rate reached 50% on the 11th day and 100% on the 39th day with a seroconversion time of 11, 12 and 14 days in median for the total antibodies, IgM and IgG.

Diagnosis of SARS-CoV-2 infection is a major public health issue. Serological tests are currently being developed. Enzyme-linked immunosorbent assay, performed on blood samples, can be performed in an automated manner and provide an estimate of the level of circulating antibody.

These serological tests could identify patients who have developed immunity to SARS-CoV-2 and be useful in the collection of epidemiological data related to COVID-19 or to know the serological status of exposed persons.

Nevertheless, SARS-CoV-2 is a new emerging virus and the antibody response (quantitative and qualitative) in COVID-19 patients is largely unknown and that of patients of HIV patients completely unknown to date. The relevance of the use of serological tests in clinical practice will indeed depend on the prior availability of physiopathological and clinical knowledge allowing their interpretation and ensuring adequate indications such as those recently proposed by the Haute Autorité de Santé ((https: //www.has -sante.fr/jcms/p_3182370/fr/premieres-indications-pour-les-tests-serologiques-du-covid-19, # 9268)).

Studies to date have shown seroconversion typically within two weeks of symptom onset, with notable differences depending on the studies, techniques and epitopes of the antigens chosen to detect the antibodies. A study which showed that the seropositivity rate reached 50% on the 11th day and 100% on the 39th day with a seroconversion time of 11, 12 and 14 days in median for the total antibodies, IgM and IgG.

Also, the immune response does not always mean protective immunization against further infection with the same virus. Only so-called neutralizing antibodies can obtain such protection. But the titer of neutralizing antibody needed to provide protection is still unknown for SARS-CoV-2. To date, the target epitopes of neutralizing antibodies have not yet been identified. In addition, data demonstrating protective immunity against COVID-19 induced by antibodies produced against SARS-CoV-2 are currently very limited.

A Chinese study that studied the antibody response in 175 patients with mild forms of COVID-19 found that 30% of them had low neutralizing antibody titer at the end of hospitalization. Differences in the titer of neutralizing antibodies were observed depending on the age of the patients, the oldest (40-59 and 60-85 years) having higher titers than the youngest (15-39 years). The titers remained stable on a control two weeks later (47/175 patients). This study raises the question of the protection of the duration of this protection.

This is why it is essential to characterize in depth the prevalence of Sars-Cov-2 infection in patients infected with HIV, patients considered to be at high risk of severe forms, and the evolution of antibody production according to the evolution of the epidemic and their protective role over time.

To date, no specific treatment or therapeutic strategy has demonstrated its effectiveness for COVID-19. Some antiretrovirals such as lopinavir / ritonavir, with in vitro activity on Sars-Cov-2, have been tested in real life with discordant results. It will be interesting to look at the antiretroviral treatments of patients who have had a Covid compared to those seronegative in serology.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* HIV + patient followed at the Pitié-Salpêtrière hospital
* Known HIV infection
* Having been informed about the study and having given oral consent (no opposition)
* Beneficiary or entitled to a social security scheme

Exclusion Criteria:

* Refusal of participation by the patient
* Patient subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective and prospective cohort study of patients infected with HIV to determine the seroprevalence of COVID-19 infection.
  This is a monocentric cohort at the Pitié-Salpêtrière hospital.
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Measure of seroprevalence of COVID-19 infection assessed by the level of anti-Covid-19 IgG antibodies in the population of people living with HIV monitored at the Pitié-Salpêtrière hospital | 12 months
  Measure of anti-SARS-CoV-2 antibodies using Abbott system

CONTACTS AND LOCATIONS:
Overall Officials: valérie Pourcher, MD, Principal Investigator — Pitie-Salpetriere Hospital
Locations (1):
- Valérie POURCHER, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No